CLINICAL TRIAL: NCT04254406
Title: 10 Years Follow-up of Patients With Residual Pockets Following the Surgical Treatment of Peri-implantitis
Brief Title: Ten Years Follow up of Peri-implant Surgery
Status: Completed | Type: Observational
Sponsor: Public Dental Service, Specialist Clinics, Sweden (Other)
Collaborators: Osaka University Japan (Unknown)
Responsible Party: Principal Investigator, Giovanni Serino, Head of Department of Periodontology, Public Dental Service, Specialist Clinics, Sweden
Other Study IDs: PDSSweden
Record Dates: First submitted 2020-01-24; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Peri-Implantitis
Keywords: Peri-Implantitis surgery; Treatment outcome; Risk factors
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Descriptive study — Evaluation of routine treatment

SUMMARY:
To report 10-years follow up of patients following the surgical treatment of peri-implantitis and to identify possible risk indicators for the progression of disease during supportive peri-implant therapy.

DETAILED DESCRIPTION:
The data for this retrospective clinical evaluation were collected from the files and radiographs of consecutive patients who had received surgical treatment of peri-implantitis between 2007 and 2009 and thereafter enrolled in supportive peri-implant treatment (SPT) .

Between 2007 and 2009, 41 patients with at least 1 implant with peri-implantitis that underwent peri-implant surgery were enrolled in a supportive peri-implant therapy.

At the 2-years follow up, two groups could be identified, one "responding group" (17 patients) who did not present any implants with peri-implantitis and a "no-responding Group" (22 patients), presenting still peri-implantitis.

Following the 2-years control visit, 17 patients of the responding group exited the supporting peri-implant therapy at the specialist clinic. They continued the routine controls at their referral clinics while the 22 patients of the no-responding group, continued the scheduled supportive peri-implant therapy (SPT) given at the specialist clinic.

ELIGIBILITY:
Inclusion Criteria:

- All patients treated with peri-implantitis surgery between 2007 and 2009 using an anti-infective protocol.

Exclusion Criteria:

* Patients treated with peri-implantitis surgery between 2007 and 2009 using a regenerative protocol at one single implants with peri-implantitis.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients who had received routine surgical treatment of peri-implantitis between 2007 and 2009 and thereafter enrolled in supportive peri-implant treatment (SPT)
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Number patients with persisting peri-implantitis following peri-implant surgery | 10 years
  The total number of patients with persisting peri-implantitis will be calculated. Any subject presenting at least one implants with a pathological pocket will be regarded as positive for the disease .
  The presence or absence of peri-implantitis will be assessed by using a periodontal probe around the mucosa of the implants.
  The definition of a pathological pocket around an implant is a pocket of 5 millimeters or more deep with concomitants bleeding after the use of the probe.
Percentage of subjects with persisting peri-implantitis | 10 years
  The percentage of patients with persisting peri-implantitis following peri-implantitis surgery will be calculated among all the patients that were treated.
  For definition of peri-implantitis see description at outcome 1.
Number of implant with persisting peri-implantitis | 10 years
  The number of implants with persisting clinical signs of peri-implantitis will be calculated. Any implant presenting a pathological pockets around its surface will be regarded as positive for the disease.
  For definition of peri-implantitis see description at outcome 1
Percentage of implants wih persisting peri-implantitis | 10 years
  The percentage of implants with persisting peri-implantitis after surgery will be calculated among all the implants that were surgically treated.
  For definition of peri-implantitis see description at outcome 1

SECONDARY OUTCOMES:
Assessement of risk factors related to the persistence of peri-implantitis | 10 years
  A univariate logistic regression to assess the correlations between each independent variable and the binary outcome presence or absence of peri-implantitis at treated implants will be used. Then, a multivariable regression analysis will be use including the independent variables from the univariate analysis that reach a statistical significance after adjusting for gender and age.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Serino, DDS PhD, Principal Investigator — Folktanvarden Specilist Clinic Periodntology
Locations (1):
- Giovanni Serino, Borås, Sweden

IPD SHARING:
Plan to Share IPD: No
After publication, on request, summary data

REFERENCES:
- [Result] Heitz-Mayfield LJA, Salvi GE, Mombelli A, Loup PJ, Heitz F, Kruger E, Lang NP. Supportive peri-implant therapy following anti-infective surgical peri-implantitis treatment: 5-year survival and success. Clin Oral Implants Res. 2018 Jan;29(1):1-6. doi: 10.1111/clr.12910. Epub 2016 Jun 23. PMID 27335316
- [Result] Serino G, Turri A, Lang NP. Maintenance therapy in patients following the surgical treatment of peri-implantitis: a 5-year follow-up study. Clin Oral Implants Res. 2015 Aug;26(8):950-956. doi: 10.1111/clr.12418. Epub 2014 May 26. PMID 24861154
- [Result] Serino G, Turri A. Outcome of surgical treatment of peri-implantitis: results from a 2-year prospective clinical study in humans. Clin Oral Implants Res. 2011 Nov;22(11):1214-20. doi: 10.1111/j.1600-0501.2010.02098.x. Epub 2011 Feb 11. PMID 21309860
- [Result] Roccuzzo M, Layton DM, Roccuzzo A, Heitz-Mayfield LJ. Clinical outcomes of peri-implantitis treatment and supportive care: A systematic review. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:331-350. doi: 10.1111/clr.13287. PMID 30328195
- [Result] Berglundh T, Armitage G, Araujo MG, Avila-Ortiz G, Blanco J, Camargo PM, Chen S, Cochran D, Derks J, Figuero E, Hammerle CHF, Heitz-Mayfield LJA, Huynh-Ba G, Iacono V, Koo KT, Lambert F, McCauley L, Quirynen M, Renvert S, Salvi GE, Schwarz F, Tarnow D, Tomasi C, Wang HL, Zitzmann N. Peri-implant diseases and conditions: Consensus report of workgroup 4 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Clin Periodontol. 2018 Jun;45 Suppl 20:S286-S291. doi: 10.1111/jcpe.12957. PMID 29926491
- [Result] Lagervall M, Jansson LE. Treatment outcome in patients with peri-implantitis in a periodontal clinic: a retrospective study. J Periodontol. 2013 Oct;84(10):1365-73. doi: 10.1902/jop.2012.120555. Epub 2012 Dec 13. PMID 23237584
- [Result] Pjetursson BE, Helbling C, Weber HP, Matuliene G, Salvi GE, Bragger U, Schmidlin K, Zwahlen M, Lang NP. Peri-implantitis susceptibility as it relates to periodontal therapy and supportive care. Clin Oral Implants Res. 2012 Jul;23(7):888-94. doi: 10.1111/j.1600-0501.2012.02474.x. Epub 2012 Apr 24. PMID 22530771